CLINICAL TRIAL: NCT04567784
Title: Neuroimaging and CBD for Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yasmin Hurd (Other)
Collaborators: GW Research Ltd (Industry)
Responsible Party: Sponsor-Investigator, Yasmin Hurd, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS#: 19-00293
Record Dates: First submitted 2020-07-30; First posted 2020-09-29 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Heroin Abuse; Opioid Use Disorder; Substance-Related Disorders; Opioid-Related Disorders
Keywords: Heroin; Opioid; Narcotics; Central Nervous System Depressants; Analgesics; Functional neuroimaging; Magnetic resonance spectroscopy
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: This study is a randomized clinical trial in which subjects will receive either placebo or 800mg cannabidiol (CBD).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants will receive a harmless, inactive solution to compare and validate the results of the other arms of the study
  Interventions: Drug: Placebo
- CBD 800mg (Experimental): Participants in Arm CBD 800 mg will receive 800mg of Cannabidiol in each of the three test sessions
  Interventions: Drug: Cannabidiol (CBD)

INTERVENTIONS:
Drug: Cannabidiol (CBD) — CBD 800 mg Cannabidiol - oral CBD solution
  Other Names: Epidiolex
  Arms: CBD 800mg
Drug: Placebo — inactive solution
  Arms: Control

SUMMARY:
The investigators propose an imaging study to investigate the neurobiological effects of CBD (vs placebo) in participants with opioid use disorder who are maintained on methadone. The purpose of the study is to determine the neural circuits and transmitters associated with the effects of CBD on to reduce craving and anxiety. The neuroimaging will be conducted in participants immediately following their first administration of CBD (800mg or placebo) and one week after the last administration (3 daily doses). This CBD administration protocol was shown in previous studies by the investigators to reduce craving and anxiety in abstinent heroin users.

DETAILED DESCRIPTION:
This study will first use multimodal imaging in individuals with opiod use disorder who are maintained on methadone to determine the neural circuits associated with the effects of CBD on craving and anxiety. Secondly, the investigators will conduct 1H MRS to characterize in-vivo neurochemical levels associated with CBD administration. Altogether, the data obtained will fill critical gaps of knowledge important in the development of a potential non-opioid medication for treating opioid use disorder.

CBD has been shown to be safe in association with opioid use and not to have severe side effects. The oral CBD solution (Epidiolex) to be used in the current study is approved by the FDA for the treatment of seizures associated with two rare and severe forms of epilepsy, Lennox-Gastaut syndrome and Dravet syndrome, in patients 2 years of age and older. Our study will investigate the neurobiological effects of CBD which is critical for its development as a potential treatment for opioid use disorder in the future. Study participation duration will last 2 weeks and will include multimodal imaging techniques to examine neural connectivity, neural activity and glutamate (and other neurometabolites) levels in relation to the impact on cue-induced responses in OUD subjects. The imagining sessions will include CBD/placebo administration; Magnetic Resonance Imaging (MRI) during task and resting-state functional MRI (rs-fMRI) and Magnetic Resonance spectroscopy (MRS); and questionnaires measuring craving, anxiety, depression, elements of cognitive function, and psychiatric history.

Screening: Study candidates will be recruited through flyers, ads and referrals from AIMS clinics. At the initial phone contact candidates will be screened for exclusion criteria and provided study information and, if they remain interested and no exclusion criteria are encountered, invited for in-person screening. Candidates will then undergo the informed consent procedure, be fully screened for eligibility and complete baseline assessments.

Randomization: Participants will be randomly assigned to either CBD or Placebo condition.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 65 years old.
* Current methadone maintenance in an opioid treatment program with a dose of =/>40mg for at least 14 days prior to participation and prescribed take-home methadone medication.
* Current opioid use disorder (OUD) or OUD in remission while on maintenance therapy with opioid agonist therapy (OAT), as determined by DSM-5 with the M.I.N.I. interview (Mini-International Neuropsychiatric Interview).
* Urinary toxicology positive for methadone.

Exclusion Criteria:

* Non-English speaking.
* Court mandate to treatment.
* Participation in another pharmacotherapeutic trial in the past 3 months.
* Poor physical health (as determined by medical screen) that would make study participation unsafe, or would prevent adherence to study procedures, including a history of cardiac disease, arrhythmias, head trauma, and seizures.
* Psychiatric conditions under DSM-5 (examined with the MINI) that would make study participation unsafe or which would prevent adherence to study procedure; examples include: suicidal or homicidal ideation requiring immediate attention, or inadequately-treated mental health disorder (e.g. active psychosis or uncontrolled bipolar disorder).
* History of impaired renal function or elevated liver enzymes >2x the normal at prescreening.
* QTc Frederica >500ms.
* Current pregnancy [determined by positive urine test] or breastfeeding.
* Not using an appropriate method of contraception such as hormonal contraception (oral hormonal contraceptives, Depo-Provera, Nuva-Ring), intrauterine device (IUD), sterilization, or double barrier method (combination of any two barrier methods used simultaneously, i.e. condom, spermicide, diaphragm).
* Medical or psychiatric contraindications for MRI (metal implants, stents, etc).
* Medical or psychiatric contraindications for CBD administration (e.g., history of hypersensitivity to cannabinoids).
* Current diagnosis of a moderate or severe substance use disorder (except for opioids and nicotine) in the past 3 months, based on DSM-5.
* Acute drug intoxication as determined by clinician assessment.
* Acute opioids withdrawal symptoms (observational and determined by the Clinical Opiate Withdrawal Scale (COWS). A Score of ≥#5 will be considered a positive result for withdrawal symptoms and/or by clinical judgment.
* Breathalyzer/Alcohol salivary/urine strips positive for alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
CBD effects on in vivo glutamatergic levels within mesocorticolimbic brain regions | 2 MRI Scans (duration 30 mins)
  Effects of CBD on in-vivo glutamatergic levels within mesocorticolimbic brain regions using Proton-Magnetic resonance spectroscopy.
Change in fMRI BOLD signal during cue reactivity | 2 MRI Scans (duration 15 mins)
  Change in fMRI blood-oxygen-level dependent (BOLD) signal acquired during the cue reactivity task at the 2nd MRI conducted 1 week after intervention as compared to the 1st MRI.
Change in fMRI BOLD signal acquired during resting-state functional connectivity | 2 MRI Scans (duration 10 mins)
  Change in fMRI blood-oxygen-level dependent (BOLD) signal acquired during resting-state at the 2nd MRI conducted 1 week after intervention as compared to the 1st MRI.

SECONDARY OUTCOMES:
Change in cue-induced drug craving on the VAS | 1 week post-intervention
  Change in cue-induced drug craving will be measured through the Visual Analogue Scale for craving, 0 (not at all) to 10 (extremely) approximately 10 days after enrollment.
Change in cue-induced anxiety on the VAS | 1 week post-intervention
  Change in cue-induced anxiety will be measured through the Visual Analogue Scale for anxiety, 0 (not at all) to 10 (extremely) approximately 10 days after enrollment.
Systolic and diastolic blood pressure (in mmHg) | 2 hours post-dose
  Change in blood pressure.
Heart rate (in beats/min) | 2 hours post-dose
  Change in heart rate.

OTHER OUTCOMES:
Adverse Events as assessed by the SAFTEE | post-intervention, approximately 1 week
  The Systematic Assessment for Treatment of Emergent Events (SAFTEE) is a structured instrument for collecting adverse drug effects.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD is not to be shared with other researchers.